Influence of volemic status on atrial natriuretic peptide in cardiac surgery patients NCT protocol 05070819

Date 15.05.2021

Objective. To identify interactions between volemic status changes and pro-ANP dynamics.

Design. Single group assessment observational open label study.

Methods. 30 cardiac surgery patients were enrolled in study. Monitoring included stroke volume variation, stroke volume, cardiac output recording (Vigileo, Edwards lifesciences). Blood samples were taken on 8 stages intraoperatively, including Teboul tests.

Statistical analysis. The normality of the distribution was estimated by the Kolmogorov–Smirnov test. The data were analyzed with a non-parametric test (Mann–Whitney U-test) to compare groups of responders and non-responders. The APACHE II and SOFA score values are presented as the mean ± standard deviation (SD). A p value ≤0.05 was considered to be statistically significant. Correlation analysis with continuous data was conducted using Pearson's correlation test (r), regression analysis. All analyses were performed using the STATISTICA data analysis software system, version 10.